CLINICAL TRIAL: NCT01202955
Title: Pilot Study of Tolcapone Effects on Abstinence-Induced Cognitive Symptoms in Smokers
Brief Title: Pilot Study of Tolcapone in Smokers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 808250
Record Dates: First submitted 2010-08-19; First posted 2010-09-16 (Estimated); Results first posted 2011-04-22 (Estimated); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Nicotine Dependence
Keywords: Smoking, Abstinence
MeSH Terms: conditions — Tobacco Use Disorder; Smoking | interventions — Tolcapone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tolcapone (Active Comparator): Tolcapone
  Interventions: Drug: Tolcapone
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tolcapone — Day 1 100mg three times per day Day 2 - Day 7 200mg three times per day Day 8 200mg twice a day Day 9 200mg once a day Day 10 100mg once a day
  Other Names: Tasmar
  Arms: Tolcapone
Drug: Placebo — Day 1 100mg three times per day Day 2 - Day 7 200mg three times per day Day 8 200mg twice a day Day 9 200mg once a day Day 10 100mg once a day
  Arms: Placebo

SUMMARY:
The goals of this within-subject pilot study are: (1) assess the feasibility and safety of administering the Catechol-O-Methyl-Transferase (COMT) inhibitor, tolcapone, to smokers, and (2) explore whether tolcapone may reduce abstinence-induced cognitive and affective symptoms that promote relapse. A secondary exploratory goal is to assess whether these effects may be more pronounced in smokers who carry a high risk COMT genotype for smoking relapse: COMT val/val.

DETAILED DESCRIPTION:
Despite decades of research to develop pharmacotherapies for nicotine dependence (ND), with current FDA approved medications (bupropion, varenicline and NRTs) the majority (>60%) of smokers relapse in the first year following treatment (Lerman, Patterson et al. 2005; Tonstad, Tonnesen et al. 2006). Testing novel medications that may reduce abstinence symptoms that prompt smoking relapse is a plausible route to identifying new treatments for nicotine dependence. The goals of this within-subject pilot study are: (1) assess the feasibility and safety of administering the Catechol-O-Methyl-Transferase (COMT) inhibitor, tolcapone, to smokers, and (2) explore whether tolcapone may reduce abstinence-induced cognitive and affective symptoms that promote relapse. A secondary exploratory goal is to assess whether these effects may be more pronounced in smokers who carry a high risk COMT genotype for smoking relapse: COMT val/val. Sixteen smokers (8 met/met genotype and 8 val/val genotype) who meet study eligibility criteria will complete two 10-day medication periods: one while taking tolcapone and one while taking placebo (order counterbalanced). The testing session will occur on day 7 of each medication phase and include three computerized tasks. Participants will be asked to refrain from smoking for at least 14 hours (overnight) prior to the testing day in each medication phase. There will be a 3-day medication taper on days 8-10 of each medication period, followed by a washout period of at least 7 days between medication periods. The main outcomes to be evaluated are participant enrollment and retention, side effects, and performance on computerized tasks. Positive results from this pilot study would provide a basis for a larger scale investigation to assess the efficacy of tolcapone as a medication that ameliorates abstinence induced neurocognitive symptoms in smokers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy as determined by a responsible physician, based on a medical evaluation including history, physical and psychiatric examination, laboratory tests, liver function monitoring.
2. Smokers who are between 18 and 55 years of age and have an IQ greater than 90.
3. Capable of giving written informed consent, which includes compliance with the requirements and restrictions, listed in the consent form.
4. Based upon self-report, subjects must smoke >10 cigarettes/day and be interested in quitting smoking in the next 6 months (i.e., treatment-seekers).
5. Women of childbearing potential must consent to using a medically accepted method of birth control (e.g., condoms and spermicide, oral contraceptive, Depo-provera injection, contraceptive patch, tubal ligation).

Exclusion Criteria:

Smoking Behavior

1. Use of chewing tobacco or snuff
2. Current enrollment or plans to enroll in another smoking cessation program in the next month
3. Plan to use other nicotine substitutes or smoking cessation treatments in the next month
4. Provide a baseline carbon monoxide (CO) reading < 10ppm

Alcohol/Drug Exclusion Criteria

1. History of substance abuse and/or currently receiving treatment for substance abuse (e.g., alcohol, opioids, cocaine, marijuana, MDMA/ecstasy, or stimulants)
2. Current alcohol consumption that exceeds >14 standard drinks/week for men and >7 standard drinks/week for women over the last 6 months

Medication Exclusion Criteria

1. Current use or recent discontinuation (within last 4-weeks) of any medication including the following:

   * Any form of psychotropic medications including:

     * antipsychotics,
     * atypical antipsychotics,
     * mood-stabilizers,
     * anti-depressants (tricyclics, SSRI's, MAOI's, nonselective MAOIs, Wellbutrin/Zyban),
     * anti-panic agents,
     * anti-obsessive agents,
     * anti-anxiety agents, and
     * stimulants (e.g., Provigil, Ritalin)
     * Varenicline
   * Medication for chronic pain
   * Anti-coagulants (e.g., Warfarin)
   * Any heart medications
   * Daily medication for asthma
   * Apomorphine, dobutamine, isoproterenol, levodopa, methyldopa, or sympathomimetic (e.g., albuterol, pseudoephedrine)
2. Current use of any smoking cessation medication.

Medical Exclusion Criteria

1. Women who are pregnant, planning a pregnancy, or lactating.
2. History or current diagnosis of psychosis, major depression or bipolar disorder, schizophrenia, or any Axis 1 disorder as identified by the MINI.
3. Serious or unstable disease within the past 6 months (e.g., cancer [except squamous cell carcinoma], heart disease, HIV, liver disease, Parkinson's disease).
4. History of epilepsy or a seizure disorder.
5. History or current diagnosis (last 6-months) of abnormal rhythms and/or tachycardia (>100 beats/minute); history or current diagnosis of chronic obstructive pulmonary disease (COPD), cardiovascular disease (stroke, angina, coronary heart disease), heart attack in the last 6 months, uncontrolled hypertension (SBP>150 or DBP>90)
6. History of Kidney and/or liver failure (including transplant) or problems (e.g., cirrhosis); current liver disease or impairment.
7. History or current diagnosis of hepatitis.
8. Liver function tests more than 20% outside of the normal range.
9. Allergies to the study medication, tolcapone (Tasmar).
10. History of severe, uncontrolled muscle movements (e.g., uncontrolled jerking, twitching) or a certain severe muscle problem (rhabdomyolysis).
11. Experience of dizziness or lightheadedness upon standing on a regular basis (i.e., daily).

Genetic Profile

1. Individuals with the heterozygous genotype (val/met) on the catechol-methyl transferase (COMT) gene. (Note: this is a small pilot study comparing effects of Tolcapone on cognitive performance between val/val (n=8) individuals.) Future research done at our center will plan to include those carrying the val/met genotype.
2. Individuals with the homozygous genotype, met/met, on the COMT gene. As of December 2008, the study has accrued 8 met/met participants. To balance the genotype groups, the study will recruit an equal number of participants with the val/val genotype on the COMT gene and not include any further participants with the homozygous, met/met genotype. Future research done at our center will plan to include those carrying the met/met genotype.
3. Non-European ancestry as determined by self report at initial telephone screening; we expect there to be ethnic differences in allele frequencies for COMT; therefore, as of December 2008, to reduce ethnic admixture that could bias the genetic analysis of this small sample, the study will be restricted to individuals of European ancestry. All participants of non-European ancestry will be referred to other studies at our center.

General Exclusion

1. Any medical condition or concomitant medication that could compromise participant safety or treatment, as determined by the Principal Investigator and/or Study Physician.
2. Inability to provide informed consent or complete any of the study tasks as determined by the Principal Investigator and/or Study Physician.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2008-07; Primary Completion 2009-05 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caryn Lerman, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited using mass media advertising from July 2008 to April 2009.
Pre-assignment Details: Each participant's catechol-o-methyl transferase (COMT) genotype was determined prior to medication assignment.
Groups:
- Tolcapone First, Then Placebo; Placebo First, Then Tolcapone: Day 1: 100mg three times per day orally Day 2 - Day 7: 200mg three times per day orally Day 8: 200mg twice a day orally Day 9: 200mg once a day orally Day 10: 100mg once a day orally
Period: Period 1: 10 Days
Arm/Group | Tolcapone First, Then Placebo | Placebo First, Then Tolcapone
Started | 9 | 10
Completed | 9 | 8
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2
Period: Period 2: 7 Days (Wash-Out)
Arm/Group | Tolcapone First, Then Placebo | Placebo First, Then Tolcapone
Started | 9 | 8
Completed | 9 | 8
Not Completed | 0 | 0
Period: Period 3: 10 Days
Arm/Group | Tolcapone First, Then Placebo | Placebo First, Then Tolcapone
Started | 9 | 8
Completed | 9 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tolcapone First, Then Placebo | Placebo First, Then Tolcapone | Total
Number analyzed (Participants) | 9 | 10 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 10 | 19
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.55 (11.41) | 40.5 (11.77) | 38.63 (11.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 3 | 6 | 9
Region of Enrollment [Number; unit: participants]
  United States | 9 | 10 | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Eligible Participants Enrolled Who Completed the Study.
Description: Number of enrolled participants who complete the final study visit
Time Frame: 30 days
Population: Number of Participants who completed the study.
Measure: Number; unit: Participants
Arm/Group | Tolcapone First, Then Placebo | Placebo First, Then Tolcapone
Number analyzed (Participants) | 9 | 10
Participants | 9 | 8

2. Secondary Outcome: N-back (Working Memory) Correct Reaction Time After Overnight Abstinence.
Description: To obtain preliminary data on the effects of Tolcapone on abstinence-induced neurocognitive deficits in abstinent smokers with differing COMT genotypes. We examined reaction time differences on the n-back task between tolcapone and placebo treatment.
Time Frame: 30 days
Population: Only participants who completed both sessions were analysed
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Tolcapone First, Then Placebo | Placebo First, Then Tolcapone
Number analyzed (Participants) | 17 | 17
Milliseconds | 597.09 (136.85) | 608.21 (151.8)

3. Secondary Outcome: Correct Reaction Time During Attention Task Performance After Overnight Abstinence.
Description: We wanted to examine the effects of Tolcapone on the Continuous Performance Task (attention task) after overnight abstinence as compared to placebo.
Time Frame: 30 days
Population: Only participants who completed both study phases were analyzed.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Tolcapone First, Then Placebo | Placebo First, Then Tolcapone
Number analyzed (Participants) | 17 | 17
Milliseconds | 460.14 (34.53) | 457.64 (39.28)

ADVERSE EVENTS:
Time Frame: 30 days
Description: No adverse events, serious or other, were reported during by any participants during this pilot study.
Groups:
- Tolcapone First, Then Placebo; Placebo First, Then Tolcapone: To maintain the study blind, both the active Tolcapone and placebo medication periods used an increased-titration dose. Below is the breakdown of the increase in dosing of the active Tolcapone:
  Day 1: 100mg three times per day orally Day 2 - Day 7: 200mg three times per day orally Day 8: 200mg twice a day orally Day 9: 200mg once a day orally Day 10: 100mg once a day orally
  During the placebo period, all participants followed the above dosing schedule; however, the capsules contained no tolcapone.
Arm/Group | Tolcapone First, Then Placebo | Placebo First, Then Tolcapone
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 0/9 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No